The Effect of Preoperative Oral Carbohydrate Administration on Postoperative Glucometabolic Response, Subjective Well Being and Quality of Life in Patients Undergoing Colorectal Surgery: A Randomized Controlled Double-Blind Study

Trial registration: NCT05402592

Date of the document: 06.03.2025

## Murat URKAN<sup>1</sup>, Cemile CELEBI<sup>2</sup>, Ulvi Mehmet MERAL<sup>3</sup>, Ikbal CAVDAR<sup>4</sup>

- <sup>1</sup> Associate Professor Doctor, Department of General Surgery, Acibadem Bodrum Hospital, Muğla, Turkey, <u>murat.urkan@acibadem.com/</u> <u>muraturkan@gmail.com</u> ORCID: 0000-0002-3191-4724
- <sup>2</sup> Assistant Professor Doctor, PhD, Muğla Sıtkı Koçman University Faculty of Health Sciences, Department of Nursing, Department of Surgical Diseases Nursing, Muğla/Turkey, cemilecelebi@mu.edu.tr/ccelebi48@gmail.com ORCID:0000-0001-9960-7205
- <sup>3</sup> Doctor, Kayseri State Hospital, Department of General Surgery, Kayseri, Turkey, ulvimeral@yahoo.com ORCID: 0000-0001-7399-6353
- <sup>4</sup> Professor Doctor, Istanbul Atlas University, Faculty of Health Sciences, Department of Nursing, Istanbul, Turkey, <a href="mailto:ikbal.cavdar@atlas.edu.tr">ikbal.cavdar@atlas.edu.tr</a> ORCID: 0000-0002-8242-6165
  - Corresponding author: Cemile ÇELEBİ/ <u>cemilecelebi@mu.edu.tr</u> /ccelebi48@gmail.com

INFORMED CONSENT FORM (For control group)

The research titled 'The effect of preoperative oral carbohydrate administration on postoperative

glucometabolic response, subjective well-being and quality of life in patients undergoing colorectal

surgery' was conducted by researchers. This research was planned to determine the effect of

preoperative fasting time on postoperative recovery. Participation in this study is voluntary. The research

will be carried out with 40 patients. Within the scope of the research, a questionnaire about your personal

information will be applied before the operation. You will be given a clear drink by your nurse to drink

at night and in the morning before the operation. On the morning of the operation, blood will be taken

from you before and 40 minutes to 90 minutes after the drink, without anaesthesia in the operating room

and the results will be evaluated. During the operation, all your vital signs will be closely monitored by

the researchers. When you are taken to your clinic after the operation, your blood sample will be taken

again at the 6th hour and 24th hour. You will be called for a follow-up by your physician on the 30th

day after your surgery. Your quality of life will be evaluated with a scale about how you spent the last

4 weeks and how much your surgery affected your life.

You can choose not to participate in the study or you can withdraw from the study even if you have

participated in the study. No sanctions will be imposed on you for this and you will not lose any of your

rights. The researchers will be able to access information about your identity, but your information will

never be disclosed even if the research is published. By signing this form, you will give permission for

people involved in the research, the organisation and the ethics committee to access your original

medical records, but this information will be kept confidential. Any information about the research topic

that may affect your continuation will be shared with you. You can contact us at ----- for anything you

wonder or want to ask during the research.

I have read all the explanations in the informed consent form. Written and verbal explanations about the

research, the subject and purpose of which are stated above, were made to me by the researcher named

below. I know that I am participating in the research voluntarily and that I can leave the research at any

time with or without justification. I agree to participate in the research with my own consent, without

any pressure or coercion.

Name-Surname of the researcher:

Name-Surname of Volunteer:

Date:

Telephone:

## INFORMED CONSENT FORM (For intervention group)

The research titled 'The effect of preoperative oral carbohydrate administration on postoperative glucometabolic response, subjective well-being and quality of life in patients undergoing colorectal surgery' was conducted by researchers. This research was planned to determine the effect of preoperative fasting time on postoperative recovery. Participation in this study is voluntary. The research will be carried out with 40 patients. Within the scope of the research, a questionnaire about your personal information will be applied before the operation. You will be given a clear drink containing carbohydrate (sugar) (12.5 g carbohydrate per 100 ml, 12% monosaccharide, 12% disaccharide, 76% polysaccharide, 285 mOsm/kg) by your nurse to drink at night and in the morning before the operation. On the morning of the operation, blood will be taken from you before and 40 minutes to 90 minutes after drinking the beverage, without anaesthesia in the operating theatre, and the results will be evaluated. During the operation, all your vital signs will be closely monitored by the researchers. When you are taken to your clinic after the operation, your blood sample will be taken again at the 6th hour and 24th hour. You will be evaluated with a scale about how you spent the last 4 weeks and how much your surgery affected your life.

You can choose not to participate in the study or you can withdraw from the study even if you have participated in the study. No sanctions will be imposed on you for this and you will not lose any of your rights. The researchers will be able to access information about your identity, but your information will never be disclosed even if the research is published. By signing this form, you will give permission for people involved in the research, the organisation and the ethics committee to access your original medical records, but this information will be kept confidential. Any information about the research topic that may affect your continuation will be shared with you. You can contact us at ----- for anything you wonder or want to ask during the research.

I have read all the explanations in the informed consent form. Written and verbal explanations about the research, the subject and purpose of which are stated above, were made to me by the researcher named below. I know that I am participating in the research voluntarily and that I can leave the research at any time with or without reason. I agree to participate in the research with my own consent, without any pressure or coercion.

| Name-Surname of the researcher: |
|---------------------------------|
| Name-Surname of the volunteer: |
| Date: |
| Telephone: |